CLINICAL TRIAL: NCT00099684
Title: A Pilot Study of the Safety, Efficacy, and Tolerability of Ezetimibe (Zetia) in Combination With Statin Therapy for the Treatment of Elevated LDL Cholesterol in HIV-Infected Subjects
Brief Title: Safety, Effectiveness, and Tolerability of Ezetimibe Combined With Statins for the Treatment of High Cholesterol in HIV Infected Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5209
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe

SUMMARY:
Anti-HIV drugs, especially protease inhibitors (PIs), have been linked to lipid metabolism problems, including elevations in low density lipoprotein cholesterol (LDL-c), triglycerides, and total cholesterol. Ezetimibe is a lipid-controlling drug; statins are part of another class of lipid-lowering drugs popularly prescribed to people with high cholesterol. The purpose of this study is to determine the safety, effectiveness, and tolerability of ezetimibe in combination with statin therapy in adults who are taking anti-HIV drugs and have high cholesterol.

Study hypothesis: In HIV infected adults, ezetimibe in combination with statin therapy will result in significantly lower LDL-c compared to statin therapy alone.

DETAILED DESCRIPTION:
Lipid metabolism abnormalities are common complications of HIV therapy, particularly with PIs. Statins and other lipid-lowering agents are often prescribed to control elevated cholesterol levels in both HIV infected and uninfected people. However, both antiretroviral therapy (ART) and lipid-lowering drugs may be associated with cardiovascular disease, so there is a clear need to find a lipid-lowering drug with low toxicity. This study will evaluate the safety, efficacy, and tolerability of ezetimibe, a lipid-controlling agent, in combination with ongoing statin therapy in HIV infected people currently on ART.

This study will last 28 weeks. All participants will be required to continue their current stable statin therapy and ART for the duration of the study.

Participants will be randomly assigned to one of two arms. Arm 1 participants will receive ezetimibe daily for 12 weeks, no treatment for 4 weeks, then placebo daily for 12 weeks. Arm 2 participants will receive placebo daily for 12 weeks, no treatment for 4 weeks, and then ezetimibe daily for 12 weeks. There will be 9 study visits; they will occur at study screening, at study entry, and every 4 weeks thereafter. Clinical assessment and blood collection will occur at all visits. Participants will be asked to complete an adherence questionnaire at Weeks 4, 12, 20, and 28, and will also be encouraged to coenroll in ACTG A5128 (Consent for Use of Stored Patient Specimens for Future Testing).

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* On ART for at least 3 months prior to study entry, and on stable ART for at least 30 days prior to study entry
* Taking one of the study-recommended statins for at least 3 months prior to study entry, and on stable statin therapy for at least 30 days immediately prior to study entry
* On lipid-lowering diet and exercise program for at least 30 days prior to screening, and willing to continue both for the duration of the study
* LDL-c of 130 mg/dL or greater within 30 days prior to study entry
* Willing to use acceptable forms of contraception
* If on hormone replacement therapy, must be on a stable dose or dose-equivalent therapy for at least 30 days prior to study entry, and must be willing to continue the same dose for the duration of the study. People taking physiologic testosterone replacement therapy are not excluded.
* If taking oral contraceptives, must be on a stable dose or dose-equivalent therapy for at least 30 days prior to study entry, and must be willing to continue the same dose for the duration of the study

Exclusion Criteria:

* Active cancer or new diagnosis of cancer within the last 5 years. People with skin cancers, including Kaposi's sarcoma, that do not require systemic treatment are not excluded.
* Prior use of ezetimibe
* Known allergy or sensitivity to ezetimibe or its components
* Diabetes mellitus or use of any diabetic medications within 30 days prior to study entry
* History of coronary heart disease
* History of or current congestive heart failure (New York Heart Association Class III or IV)
* Known atherosclerotic disease risk (e.g., history of myocardial infection, bypass surgery, angioplasty, angina pectoris with a positive stress test or angiographic documentation)
* Vascular abnormalities (e.g., cerebrovascular disease, peripheral vascular disease, abdominal aortic aneurysm, or leg artery blockages)
* Untreated or uncontrolled hypothyroidism
* Current drug or alcohol abuse that may interfere with the study
* Testosterone therapy beyond normal physiologic levels of the hormone within 3 months prior to study entry
* Initiation or change in physiologic testosterone replacement therapy within 3 months prior to study entry
* Hormonal anabolic therapies within 3 months prior to study entry
* Systemic cancer chemotherapy or immunomodulators (e.g., growth factors, immune globulin, interleukins, and interferons) within 60 days prior to study entry
* Lipid-lowering agents (except statins) within 30 days prior to study entry
* Any corticosteroid therapy above replacement levels within 30 days prior to study entry
* Untreated or uncontrolled hypertension
* Active AIDS-defining opportunistic infection (OI) within 30 days prior to study entry. People who have no evidence of active disease and are receiving maintenance therapy for AIDS-related OIs are not excluded.
* Acute illness that would interfere with the study within 30 days prior to study entry
* Investigational agents. People using expanded access investigational antiretroviral drugs are not excluded.
* Decreased mental capacity that may interfere with the study
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-11; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change in directly measured fasting LDL-c while receiving ezetimibe compared to change while receiving placebo
changes in clinical symptoms and safety labs while receiving ezetimibe compared to changes in clinical symptoms while receiving placebo

CONTACTS AND LOCATIONS:
Overall Officials: Susan Koletar, MD, Study Chair — Division of Infectious Diseases, Ohio State University; Dominic Chow, MD, MPH, Study Chair — University of Hawaii, Hawaii AIDS Clinical Research Program, Leahi Hospital
Locations (42):
- United States (41):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA School of Medicine, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - University of California, San Diego Antiviral Research Center, San Diego, California
  - San Francisco General Hospital, San Francisco, California
  - San Mateo County AIDS Program, Stanford, California
  - Santa Clara Valley Medical Center, Stanford, California
  - Stanford University, Stanford, California
  - Willow Clinic, Stanford, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - University of Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian/St. Lukes (Chicago), Chicago, Illinois
  - Cook County Hospital Core Center, Chicago, Illinois
  - Feinberg School of Medicine, HIV/ACTU, Chicago, 60611-3015, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Wishard Hospital, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Nebraska Health System, Omaha, Nebraska
  - SUNY - Buffalo (Rochester), Buffalo, New York
  - Beth Israel Medical Center, New York, New York
  - Chelsea Clinic, New York, New York
  - NYU/Bellevue, New York, New York
  - The Cornell Clinical Trials Unit, New York, New York
  - Columbia University, New York, New York
  - Community Health Network, Inc., Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Presbyterian Medical Center - Univ. of PA, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Stanley Street Treatment and Resource, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Comprehensive Care Clinic, Nashville, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - University of Texas, Galveston, Galveston, Texas
  - University of Washington (Seattle), Seattle, Washington
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Calza L, Manfredi R, Chiodo F. Dyslipidaemia associated with antiretroviral therapy in HIV-infected patients. J Antimicrob Chemother. 2004 Jan;53(1):10-4. doi: 10.1093/jac/dkh013. Epub 2003 Nov 25. PMID 14645323
- [Background] Colagreco JP. Cardiovascular considerations in patients treated with HIV protease inhibitors. J Assoc Nurses AIDS Care. 2004 Jan-Feb;15(1):30-41. doi: 10.1177/1055329003256922. PMID 14983559
- [Background] Martinez E, Tuset M, Milinkovic A, Miro JM, Gatell JM. Management of dyslipidaemia in HIV-infected patients receiving antiretroviral therapy. Antivir Ther. 2004 Oct;9(5):649-63. PMID 15535403
- [Background] Visnegarwala F, Maldonado M, Sajja P, Minihan JL, Rodriguez-Barradas MC, Ong O, Lahart CJ, Hasan MQ, Balasubramanyam A, White AC Jr. Lipid lowering effects of statins and fibrates in the management of HIV dyslipidemias associated with antiretroviral therapy in HIV clinical practice. J Infect. 2004 Nov;49(4):283-90. doi: 10.1016/j.jinf.2003.09.006. PMID 15474625
- See also: Click here for more information about ACTG A5128 — http://clinicaltrials.gov/ct/show/NCT00031408